CLINICAL TRIAL: NCT04436887
Title: Prophylactic Sub-lay Non-absorbable Mesh Following Emergent Midline Laparotomy Clean/Contaminated Field: Early Results of a Randomized Double-blind Prospective Trial: PROMETHEUS
Brief Title: Prophylactic Sub-lay Non-absorbable Mesh Following Midline Laparotomy: PROMETHEUS (PROphylactic Mesh Trial Evaluation UltraSound)
Acronym: PROMETHEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francesco Pizza (Other)
Responsible Party: Sponsor-Investigator, Francesco Pizza, Head of bariatric unit, Azienda Sanitaria Locale Napoli 2 Nord
Organization: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 11062018
Record Dates: First submitted 2020-06-13; First posted 2020-06-18 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Incisional Hernia; Wound Infection
MeSH Terms: conditions — Incisional Hernia; Wound Infection

STUDY DESIGN:
Intervention Model Description: Sample size: Considering a mean percentage of incidence of Incisional Hernia of 20% in the open middle line laparotomy in the clean-contemned setting. We hypothesized that Incisional Hernia rate in Group B (Experimental Group) would be superior to Group A (control group) if the difference in a mean percentage of incidence of Incisional Hernia was less than 15%. 194 patients are required to have a 90% chance of detecting, as significant at the 5% level, a decrease in the primary outcome measure from 20% in the control group to 5% in the experimental group. Baseline comparisons were performed using chi-square tests and T-tests. Continuous variables are expressed as mean ± standard deviation (SD). Differences between preoperative and postoperative parameters were compared by Wilcoxon paired rank test. For all tests, a two-sided p<0.05 was considered statistically significant. The study designed with Sealed Envelope.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding Process
  Patients, care providers, staff collecting data, and those assessing the endpoints were all blinded to treatment allocation. Patients were blinded to the surgical procedure performed until the final assessment of the study endpoints. Because the blinding of the operating surgeons was not feasible, they were not involved in the data collection and outcome assessment. Physicians in charge of patients' management were not involved in the operating room and were blinded to the intervention. The data were collected and analyzed by physicians who were not involved in the patient's management during the whole Randomized Controlled Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Primary closure (No Intervention): Primary closure of midline laparotomy
- Mesh closure (Experimental): Sub-lay permanent mesh supported the closure
  Interventions: Procedure: positioning of polypropylene strips for prophylactic purposes in closing the middle laparotomies to prevent the incisional hernia

INTERVENTIONS:
Procedure: positioning of polypropylene strips for prophylactic purposes in closing the middle laparotomies to prevent the incisional hernia — Sub-lay mesh supported closure A 4 cm space is created between posterior rectus sheath and rectus muscle, widening 2 cm at each side of midline. Both posterior rectus sheath edges are sutured using a running slowly absorbable suture. Above arcuate line, posterior layer was performed suturing peritoneum and posterior rectus sheath; below arcuate line, posterior layer was performed suturing peritoneum and trasversalis fascia. Anterior layer was performed suturing anterior rectus sheath. A suture length to wound length ratio of 4:1 is recommended. A 4-cm Parietex Progrip Mesh strip was placed between the posterior rectus sheath and rectus muscle with an overlap of at least 2 cm at each side, suture less. In laparotomies >20 cm two stripes of 15 cm each were designed. The midline anterior rectus sheath was closed using a running slowly absorbable suture, covering the mesh. A suture length to wound length ratio of 4:1 is recommended.
  Arms: Mesh closure

SUMMARY:
The aim of the present study is to analyse feasibility, safety and Incisional Hernia rate using a prophylactic sub lay non-absorbable mesh [Parietex Progrip (Medtronic) ] in order to prevent Incisional Hernia following midline emergent laparotomy in clean and clean-contaminated wounds.

DETAILED DESCRIPTION:
The study is a double-blinded randomized trial, comparing the widely recommended midline laparotomy closure using a running slowly absorbable suture to closure with the aid of a permanent sub-lay mesh (Parietex Progrip), in patients undergoing midline laparotomy for clean-contaminated surgery. From January 2016 to June 2018, a series of 200 patients were included. All patients were operated in a single surgical Unit, located in Lacco Ameno (Naples) at the only Hospital of the island. All patients undergoing 'open' midline laparotomy for abdominal surgery in clean-contaminated fields were included. All patients subscribed informed consent. Authorization was requested from the local regional Ethics Committee. Exclusion criteria were: age < 18 years; life expectancy < 24 months (as estimated by the operating surgeon), pregnancy, immunosuppressant therapy within 2 weeks before surgery, clean, contaminated and dirty wounds, wound length<10 cm. Patients were randomized in two groups (Group A, receiving primary closure; Group B, receiving mesh supported closure in a Sublay fashion). Randomization was obtained just before abdominal wall closure through number (1 to 200) extraction by Operative room nurse (Even: Group A vs Odd: Group B). All patients enrolled in the study were followed up sending a letter to their General Practitioner. Outpatient clinic controls were done by surgeons/surgical residents/General Practitioner blinded for the procedure.

Technical details Group A. Primary closure of midline laparotomy. The midline fascia is closed using a double layer running slowly absorbable suture. Above arcuate line, the posterior layer was performed suturing peritoneum and posterior rectus sheath; below arcuate line posterior layer was performed suturing peritoneum and trasversalis fascia. Anterior layer was performed suturing anterior rectus sheath. Suture length to wound length ratio of 4:1 as recommended (not routinely measured). Subcutaneous tissue and skin are closed according to the first surgeon's preference.

Group B. Sub-lay mesh supported closure A 4 cm space is created between posterior rectus sheath and rectus muscle, widening 2 cm at each side of midline. Both posterior rectus sheath edges are sutured using a running slowly absorbable suture. Above the arcuate line, the posterior layer was performed suturing peritoneum and posterior rectus sheath; below the arcuate line, the posterior layer was performed suturing peritoneum and trasversalis fascia. The anterior layer was performed suturing anterior rectus sheath. A suture length to wound length ratio of 4:1 is recommended (not routinely measured). A 4-cm Parietex Progrip Mesh strip was placed between the posterior rectus sheath and rectus muscle with an overlap of at least 2 cm at each side, sutureless. The not gripping face of the mesh was positioned on the posterior rectal sheat to allow the muscle to become in contact with the grips. In laparotomies >20 cm two stripes of 15 cm each were designed. The midline anterior rectus sheath was closed using a running slowly absorbable suture covering the mesh. A suture length to wound length ratio of 4:1 is recommended (not routinely measured). Subcutaneous tissue and skin closure were up to the surgeon preference.

Endpoints Primary endpoint was Incisional Hernia rate. Patients were postoperatively examined at 3, 6, 12 and 24 months. Both clinical examination and ultrasound imaging were performed in all patients at follow-up. Physicians were blind about which Group (A or B) the patients had been placed. Incisional Hernia was clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar. At 3, 6, 12 and 24 months ultrasound imaging was performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia were registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia were a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia was diagnosed if clinical criteria and/or ultrasound criteria were fulfilled. The study was not designed to discriminate single or multiple defects. The study will be completed at 2 years' follow up. Secondary endpoints included the incidence of wound events. Wound events were classified as surgical site infections according to Clavien Dindo criteria (superficial, deep or organ space). Surgical site events were reported according to the Ventral Hernia Working Group definitions. Actions for wound events were categorized as follows: antibiotics only, bedside wound interventions, percutaneous manoeuvres or surgical debridement.

Blinding Process

Patients, care providers, staff collecting data, and those assessing the endpoints were all blinded to treatment allocation. Patients were blinded to the surgical procedure performed until the final assessment of the study endpoints. Because the blinding of the operating surgeons was not feasible, they were not involved in the data collection and outcome assessment. Physicians in charge of patients' management were not involved in the operating room and were blinded to the intervention. The data were collected and analyzed by physicians who were not involved in the patient's management during the whole Randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Clean-contaminated wounds
* midline laparotomy >10 cm
* Informed consent

Exclusion Criteria:

* age < 18 years;
* life expectancy < 24 months (as estimated by the operating surgeon), -
* pregnancy
* immunosuppressant therapy within 2 weeks before surgery
* clean, contaminated and dirty wounds
* wound length<10 cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 3 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 6 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 12 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar
Rate of Incisional Hernia at Clinical examination | Patients are postoperatively examined at 24 months.
  Clinical examination: Incisional Hernia is clinically defined as any visible or palpable ''blowout'' in the midline abdominal scar.
Rate of Incisional Hernia at Ultrasound examination | Patients are postoperatively examined at 3 months.
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.
Rate of Incisional Hernia at Ultrasound examination | Patients are postoperatively examined at 6 months.
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.
Rate of Incisional Hernia at Ultrasound examination | Patients are postoperatively examined at 12 months.
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.
Rate of Incisional Hernia at Ultrasound examination | Patients are postoperatively examined at 24 months.
  Ultrasound imaging is performed to examine the midline for all patients with symptomatic or asymptomatic, providing any valuable information about Incisional Hernia onset. Size and location of all ultrasound detected Incisional Hernia are registered, as well as any other patient's complaint. The ultrasonic criteria of Incisional Hernia are a visible gap within the abdominal wall and/or ''tissue moving through the abdominal wall by Valsalva manoeuvre'' and/or a detectable ''blowout''. Incisional Hernia is diagnosed if clinical criteria and/or ultrasound criteria are fulfilled.

SECONDARY OUTCOMES:
Number of patients affected by Superficial surgical site infections | Within 30 days postoperatively
  Superficial infections according to Clavien-Dindo criteria
Number of patients affected by Deep surgical site infections | Within 30 days postoperatively
  Deep surgical site infections according to Clavien-Dindo criteria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pizza F, D'Antonio D, Lucido FS, Del Rio P, Dell'Isola C, Brusciano L, Tolone S, Docimo L, Gambardella C. Is absorbable mesh useful in preventing parastomal hernia after emergency surgery? The PARTHENOPE study. Hernia. 2022 Apr;26(2):507-516. doi: 10.1007/s10029-022-02579-w. Epub 2022 Feb 23. PMID 35195798
- [Derived] Pizza F, D'Antonio D, Ronchi A, Lucido FS, Brusciano L, Marvaso A, Dell'Isola C, Gambardella C. Prophylactic sublay non-absorbable mesh positioning following midline laparotomy in a clean-contaminated field: randomized clinical trial (PROMETHEUS). Br J Surg. 2021 Jun 22;108(6):638-643. doi: 10.1093/bjs/znab068. PMID 33907800